CLINICAL TRIAL: NCT03189537
Title: Double Blind Randomised Placebo Controlled Trial for Evaluation of Efficacy and Safety of Ingavirin® for Post-exposure Profilaxis During Rise in the Incidence of Influenza and Other Acute Respiratory Viral Infections in Adults
Brief Title: Study of Post-Exposure Ingavirin® Prophylaxis of Influenza and Acute Respiratory Viral Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2P/09
Record Dates: First submitted 2017-06-08; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Influenza, Human; Acute Respiratory Infection; Common Cold; Flu; Viral Infection
Keywords: Profilaxis; Ingavirin
MeSH Terms: conditions — Influenza, Human; Common Cold; Virus Diseases | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin (Experimental): Ingavirin (Imidazolyl Ethanamide Pentandioic Acid) capsules, 90 mg once daily for 7 days
  Interventions: Drug: Ingavirin (Imidazolyl Ethanamide Pentandioic Acid)
- Placebo (Placebo Comparator): Placebo oral capsule, once daily for 7 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ingavirin (Imidazolyl Ethanamide Pentandioic Acid) — Broad-spectrum antiviral agent
  Arms: Ingavirin
Drug: Placebo oral capsule — Placebo capsule to match Ingavirin capsule
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate efficacy of prophylactic Ingavirin intake by people having contact with sick people infected with influenza and other acute respiratory viral infections

DETAILED DESCRIPTION:
The study includes 7 days of treatment period and 30 days of follow-up, 37 days total.

The participant was receiving Ingavirin or placebo for 7 days. Then during 30 days the participant was under supervision.

Visits were performed at days 2-7 (every day) since inclusion and then every 5 days during follow-up period.

Wherever during the study the participant developed symptoms of flu or other acute respiratory viral infection, the participant was taken for medical care to observe his condition, symptoms dynamics, lab tests, including laboratory verification of viral origin of the disease. Medical care was established for 10±2 days since symptoms. Everyday for 3 days and additional visits for 5±1 and 10±2 days of the disease.

The patient had the required symptomatic treatment, additionally the patient could be institutionalised if necessary.

Wherever the participant developed symptoms during treatment period, the patient was taken investigational drug on schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participants who do have continuous contact with ill person (staff members, dormitory, family members), laboratory confirmed viral origin, during influenza/other acute viral respiratory disease season
* First exposure with the ill person who is present with symptoms of flu or acute respiratory viral infection (fever, intoxication, catarrhal symptoms) ≤ 48 hours
* Signed Informed Contest to participate in the study
* Contraception throughout the study

Exclusion Criteria:

* Interferone or interferone inducers intake, or substances with action on immune system intake less then 3 months before inclusion
* Anti-virals intake, other then investigational drug, throughout the study
* Vaccination for Influenza less than 1 year before inclusion
* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-10-03 (Actual); Primary Completion 2011-04-19 (Actual); Study Completion 2011-10-10 (Actual)

PRIMARY OUTCOMES:
Difference in incidence of flu / other acute respiratory viral infections between Ingavirin and placebo groups | Through study completion, an average of 37 days
  To evaluate incidence difference between Ingavirin and placebo groups. Incidence defined as ratio between number of people got sick in the group to all people in the group. 1) Efficiency Index (EI) was defined as incidence of flu in placebo group to incidence of flu in Ingavirin group. 2) Efficacy Ratio (ER) defined by formula: ER=(incidence in placebo group - incidence Ingavirin group)*100% then divided by incidence in placebo group.

SECONDARY OUTCOMES:
Comparative evaluation of prevalence and duration of flu and acute viral respiratory infection at participants who developed flu / avri | Through study completion, an average of 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Zakharova, MD, PhD, Study Director — Valenta Pharm JSC
Locations (2):
- Russia (2):
  - Research Institute of Influenza, Saint Petersburg
  - Saratov State Medical University named after V. I. Razumovsky, Saratov

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shul'diakov AA, Liapina EP, Kuznetsov VI. [Current principles in the chemoprophylaxis of acute respiratory viral infections]. Ter Arkh. 2013;85(11):27-33. Russian. PMID 24432596